CLINICAL TRIAL: NCT01110590
Title: Randomized, Double-blind, Placebo-controlled, Group-comparison, Dose-escalation Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Co-administration of Different Doses of Vardenafil (2 Dose Strengths) and BAY60-4552 (4 Dose Strengths) Given Once-daily (od) Over 14 Days in Patients With Erectile Dysfunction (ED).
Brief Title: Multiple Dose Escalation Study (14 Days) to Investigate Safety, Tolerability, PK and PD of Vardenafil and BAY60-4552
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Head Clinical Pharmacology, Bayer HealthCare AG
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 14612; 2009-015894-11 (EudraCT Number)
Record Dates: First submitted 2010-04-14; First posted 2010-04-26 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — BAY 60-4552; Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: BAY60-4552 + Vardenafil
- Arm 2 (Experimental)
  Interventions: Drug: BAY60-4552 + Vardenafil
- Arm 3 (Experimental)
  Interventions: Drug: BAY60-4552 + Vardenafil
- Arm 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BAY60-4552 + Vardenafil — Total dose given over 14 days: 5.25 mg BAY60-4552 + 140 mg Vardenafil
  Arms: Arm 1
Drug: BAY60-4552 + Vardenafil — Total dose given over 14 days: 21.0 mg BAY60-4552 + 140 mg Vardenafil
  Arms: Arm 2
Drug: BAY60-4552 + Vardenafil — Total dose given over 14 days: 21.0 mg BAY60-4552 + 280 mg Vardenafil
  Arms: Arm 3
Drug: Placebo — Placebo
  Arms: Arm 4

SUMMARY:
Safety, tolerability, pharmacokinetics and pharmacodynamics will be investigated in this multiple dose escalation study. In three treatments groups different dosages of BAY 60-4552 and vardenafil will be given with patients with erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* The informed consent must be signed before any study specific tests or procedures are done
* Male patients with a history of erectile dysfunction (ED) for at least 6 months, defined as "the inability to achieve and maintain an erection of the penis sufficient to complete satisfactory sexual intercourse" by the NIH consensus report 1993. The diagnosis of 'Erectile dysfunction' has to be confirmed by a physician
* Age: 18 to 70 years (inclusive) at the first screening examination
* Ethnicity: White
* Body mass index (BMI): equal to or above 18 and below 32 kg / m²
* Confirmation of the patient's health insurance coverage prior to the first screening examination / visit
* Ability to understand and follow study-related instructions

Exclusion Criteria:

* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal
* Known hypersensitivity to the study drugs (active substances or excipients of the preparations)
* Known severe allergies, non-allergic drug reactions, or multiple drug allergies
* Any underlying cardiovascular condition, including unstable angina pectoris that would preclude sexual activity according to the NIH consensus report 1993
* History of myocardial infarction, stroke or life-threatening arrhythmia within 6 months prior to screening
* Bleeding disorder
* History of prostatectomy because of prostate cancer, including nerve-sparing techniques. Clarification: Any surgical procedures for the treatment of Benign Prostate Hypertrophy (BPH) are permitted, with the exception of cryosurgery, cryotherapy or cryoablation
* Hereditary degenerative retinal disorders such as retinitis pigmentosa
* History of loss of vision because of NAION (Bayer Study 12912), temporary or permanent loss of vision, including unilateral loss of vision
* History of uni- or bilateral hearing loss

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Adverse Event reporting | up to 6 weeks

SECONDARY OUTCOMES:
Plasma concentration of study drugs; Pharmacokinetic parameters: AUC, Cmax, AUC/D, Cmax;norm, Cmax/D, t1/2, tmax | Day 0, 6, 13
Plasma concentration of cyclic guanosine monophosphate (cGMP) | Day 0, 6, 13

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Mönchengladbach, North Rhine-Westphalia, Germany